CLINICAL TRIAL: NCT04375540
Title: Vertical Gingival Display Changes Associated With Upper Premolars Extraction Orthodontic Treatment in Gummy Smile Patients: A Prospective Clinical Trial
Brief Title: Vertical Gingival Display Changes Associated With Upper Premolars Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Elham Abu Alhaija, Professor, Jordan University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 285/2016
Record Dates: First submitted 2020-05-02; First posted 2020-05-05 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Gummy Smile; Orthodontic Treatment
Keywords: Gingival display; Tooth extraction; Dental esthetics; Corrective orthodontics

STUDY DESIGN:
Intervention Model Description: Group 1: upper first premolars extraction (24 patients) Group 2: upper second premolars extraction (26 patients) and Group 3: no orthodontic intervention was performed (happy with their teeth) (26 subjects).
Who Masked: Outcomes Assessor
Masking Description: Study casts and cephalometric analysis were performed by different person (D. T.) who did not know to which group the patient belongs. Records were given numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Upper first premolars extraction (Experimental): Included 24 patients (7 males,17 females) with a mean age of 21.56±3.19years who were treated with fixed orthodontic appliance for 2.22±0.31years.
  Interventions: Procedure: Upper first premolars extractions
- Upper second premolars extraction (Experimental): Included 26 patients (8 males,18 females) with a mean age of 22.16±3.59years who were treated with fixed orthodontic appliance for 2.25±0.30 years.
  Interventions: Procedure: Upper second premolars extraction
- No intervention (No Intervention): Included 26 subjects (10 males, 16 females) with a mean age of 20.45±3.29years.This group was included to observe any changes in the vertical gingival display over the 2 years' observation period (1.65±0.17 years).

INTERVENTIONS:
Procedure: Upper first premolars extractions — Fixed orthodontic treatment with upper first premolars extraction and space closure using 0.019X0.025 SS AW and elastic chain.
  Arms: Upper first premolars extraction
Procedure: Upper second premolars extraction — Fixed orthodontic treatment with upper second premolars extraction and space closure using 0.019X0.025 SS AW and elastic chain.
  Arms: Upper second premolars extraction

SUMMARY:
To investigate and compare vertical gingival display (VGD) changes associated with upper premolars extraction during orthodontic treatment.

DETAILED DESCRIPTION:
Seventy-six subjects who met the inclusion criteria were divided into one of 3 groups according to their treatment modalities as follows: group 1: upper first premolars extraction (24 patients, aged 21.56±3.19 years); group 2: upper second premolars extraction (26 patients, aged 22.16±3.59 years) and group 3: no orthodontic intervention was performed (happy with their teeth) (26 subjects, aged 20.45±3.29 years).

Initial records (radiographs, study casts and clinical photographs) were taken for all subjects. The same records were taken post treatment for treated subjects only. The Pre- and post- treatment VGD and lip length in static and dynamic positions and the amount of upper teeth retractions were recorded.

The paired t-test and ANOVA test were used to detect treatment changes and differences between studied groups, respectively. Factors affecting VGD were investigated using backward stepwise linear regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* age 17 years or more
* skeletal class I or class II malocclusion
* upper premolars extraction treatment plan
* high smile line 2mm or more
* no previous orthodontic treatment.

Exclusion Criteria:

* poor oral hygiene
* lower arch extraction treatment plan
* smoking
* Any systemic or periodiontal disease.

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
The amount of pre- and post-treatment vertical gingival display in static and dynamic positions. | 2 years
  Measured from the lower edge of the upper lip to the gingival margins of the incisors in mm.
Pre- and post treatment Nose-U-lip-length | 2 years
  Measured from the soft tissue subnasale to the upper lip stomion (base of the nose to the lip edge of the upper lip) in mm.
Upper anterior teeth retraction | 2 years
  The amount of upper anterior teeth edges' retraction on cephalometric superimposition in mm
Upper incisors extrusion | 2 years
  The amount of upper incisors edges vertical displacement on cephalometric superimposition in mm

SECONDARY OUTCOMES:
Upper molars protraction | 2 years
  The amount of upper molars protraction measured from the mesial contact point of the molar in the baseline model to the mesial contact point of the transposed transparent model(S1) in mm

CONTACTS AND LOCATIONS:
Overall Officials: Elham Abu Alhaija, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Faculty of Dentistry/ Jordan university of Science and Technology Dental Teaching cliniucs, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No